CLINICAL TRIAL: NCT02134457
Title: Multicenter Randomized Double Masked Parallel Design Exploratory Study to Assess Safety and Efficacy of Two Different Doses of Intravitreal Anti-VEGF Treatment With Ranibizumab (0.12 mg vs. 0.20 mg) in Infants With Retinopathy of Prematurity (ROP)
Brief Title: Comparing Alternative Ranibizumab Dosages for Safety and Efficacy in Retinopathy of Prematurity
Acronym: CARE-ROP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Andreas Stahl, MD, MD, University Hospital Freiburg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CARE-ROP; 2013-002539-13 (EudraCT Number)
Record Dates: First submitted 2014-04-26; First posted 2014-05-09 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Retinopathy of Prematurity (ROP)
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranibizumab 0.12 mg (Experimental): 20 µl of the 6 mg/ml ranibizumab concentration will be applied intravitreally. After an initial response the same dose as in the first injection can be re-applied after at least four weeks post injection.
  A maximum number of 3 regular re-injections can be applied.
  Interventions: Biological: ranibizumab
- Ranibizumab 0.20 mg (Experimental): 20 µl of the 10 mg/ml ranibizumab concentration will be applied intravitreally. After an initial response the same dose as in the first injection can be re-applied after at least four weeks post injection.
  A maximum number of 3 re-injections can be applied.
  Interventions: Biological: ranibizumab

INTERVENTIONS:
Biological: ranibizumab
  Other Names: Lucentis

SUMMARY:
This study is designed as an exploratory study to assess safety and efficacy of two different doses of the anti-VEGF agent ranibizumab (0.12 mg vs. 0.20 mg) in the treatment of infants with retinopathy of prematurity. Furthermore it shall help to improve safety in the treatment of ROP and provide explorative data on long-term effects of ranibizumab after intravitreal injection in neonates.

The primary objective is to assess clinical efficacy of ranibizumab in children with ROP

ELIGIBILITY:
Inclusion Criteria:

* Bilateral ROP in zone I (stage 1+, 2+, 3+/-, AP-ROP) or ROP in central (=posterior) zone II (stage 3+, AP-ROP). Zone I is defined as twice the distance from the optic disc to the fovea measured temporally, posterior zone II is defined as three times the distance from the optic disc to the fovea measured temporally.
* Legal representatives or their designates willing and able to attend regular study visits with the study infant.
* Written informed consent to participate in the study (signed by all patient's legal representatives).

Exclusion Criteria:

* Pediatric conditions rendering the infant ineligible to anti-VEGF treatment or to repeated blood draws as evaluated by a neonatal ICU specialist and a study ophthalmologist.
* Congenital brain lesions significantly impairing optic nerve function.
* Severe hydrocephalus with significantly increased intracranial pressure.
* Advanced stages of ROP with partial or complete retinal detachment (ROP stage 4 and 5).
* ROP involving only the peripheral retina (i.e. peripheral zone II or zone III).
* Known hypersensitivity to the study drug or to drugs with similar chemical structures.
* Contraindications for an intravitreal injection as listed in ranibizumab SmPC.
* Systemic use of anti-VEGF therapeutics.
* Use of other investigational drugs - excluding vitamins and minerals - at the time of enrollment, or within 30 days or 5 half-lives prior to enrollment, whichever is longer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-08; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment | Up to 24 weeks post first injection
  Efficacy is determined by the number of infants without need for rescue treatment up to week 24 post first injection.
  Re-injection of study dose is not considered rescue treatment if applied after an initial response to treatment and after at least 4 weeks post injection.

SECONDARY OUTCOMES:
Regression of plus disease | Up to 24 weeks post first injection
Regression of preretinal vascularized ridge | Up to 24 weeks post first injection
Progression of peripheral intraretinal vascularization beyond ridge | Up to 24 weeks post first injection
Number and kind of AEs and SAEs | Up to 24 weeks post first injection
Changes in vascular endothelial growth factor (VEGF) levels in the systemic circulation | Up to 24 weeks post first injection
Number of re-injections of study dose | Up to 24 weeks post first injection
Number of patients progressing to stage 4 or 5 ROP | Up to 24 weeks post first injection
Number of patients with complete vascularization of the peripheral retina to within one disc diameter of the ora serrata | Up to 24 weeks post first injection

OTHER OUTCOMES:
Number of late recurrences of ROP during the follow-up period | Up to 5 years post first injection
Number of patients progressing to stage 4 or 5 ROP after the core study | Up to 5 years post first injection
Number of patients with complete vascularization of the peripheral retina to within one disc diameter of the ora serrata after the end of the core study | Up to 5 years post first injection
Long-term ophthalmological development: visual acuity (if possible), orthoptic status, cycloplegic retinoscopy, refraction, IOP, fundoscopy including fundus photographs | Up to 5 years post first injection
  At one year and at 5 years an ophthalmological visit will take place.
Long-term pediatric development: Bayley-test, weight, height, cognitive, motor and sensory development | Up to 5 years post first injection
Number and kind of AEs or SAEs per group between the end of the observational core study and the end of the follow-up period | Up to 5 years post first injection

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Stahl, MD, Principal Investigator — University Eye Hospital Freiburg, Germany
Locations (9):
- Germany (9):
  - University Eye Hospital, Freiburg im Breisgau, Baden-Wurttemberg
  - University Eye Hospital, Bonn
  - University Eye Hospital, Düsseldorf
  - University Eye Hospital, Kiel
  - University Eye Hospital, Magdeburg
  - University Eye Hospital, Munich
  - University Eye Hospital, Münster
  - University Eye Hospital, Regensburg
  - University Eye Hospital, Tübingen

REFERENCES:
- [Derived] Stahl A, Krohne TU, Eter N, Oberacher-Velten I, Guthoff R, Meltendorf S, Ehrt O, Aisenbrey S, Roider J, Gerding H, Jandeck C, Smith LEH, Walz JM; Comparing Alternative Ranibizumab Dosages for Safety and Efficacy in Retinopathy of Prematurity (CARE-ROP) Study Group. Comparing Alternative Ranibizumab Dosages for Safety and Efficacy in Retinopathy of Prematurity: A Randomized Clinical Trial. JAMA Pediatr. 2018 Mar 1;172(3):278-286. doi: 10.1001/jamapediatrics.2017.4838. PMID 29309486